CLINICAL TRIAL: NCT06869616
Title: CRacking the HEterogeneity of Social Outcome Through Neuropsychophysiological Profiles
Acronym: CRHESO
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Giulia Agostoni, PsyD, PhD, IRCCS San Raffaele
Other Study IDs: CRHESO
Record Dates: First submitted 2025-02-28; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Schizophenia Disorder
Keywords: electrophysiology; metaphor comprehension; language disorder; social functioning
MeSH Terms: conditions — Language Disorders; Social Adjustment | interventions — Cognitive Remediation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Schizophrenia Group: We will enroll 50 patients selected according to the presence of Schizophrenia diagnosis (DSM V criteria), which will be tested for metaphor comprehension, as well as for the other variables included in the study, and the electrical brain activity will be registered through a 128 channel EEG.
  Among these, a subgroup of 10 subjects will undergo a cognitive remediation training (Cognitive Remediation), already published and demonstrated to be feasible for patients with schizophrenia. Specifically, it consists of 15 sessions of 45 minutes each, including computerized domain-specific neurocognitive exercises aimed at training specific cognitive areas known to be impaired in schizophrenia.
  Interventions: Other: Cognitive Remediation
- Healthy controls: 50 healthy subjects, as control sample, that will be tested for metaphor comprehension, as well as for the other variables included in the study, and the electrical brain activity will be registered through a 128 channel EEG.

INTERVENTIONS:
Other: Cognitive Remediation — 10 patients will undergo a rehabilitative training (Cognitive Remediation), already published and demonstrated to be feasible for patients with schizophrenia. This program includes domain-specific neurocognitive exercises aimed at training specific cognitive areas known to be impaired in schizophrenia. The treatment plan includes 15 45-minutes sessions.
  Groups: Schizophrenia Group

SUMMARY:
CRHESO aims at overcoming the considerable burden of mental disorders, which affects both psychosocial well-being and societal welfare, through a multidisciplinary and integrated approach to explore and remediate dimensions affecting social outcome.

DETAILED DESCRIPTION:
Social functioning is fundamental for human adaptation, relationships, and psychological well-being. Schizophrenia, a severe psychiatric disorder, is one of the leading causes of disability worldwide and presents significant challenges in social interactions for those affected, increasing the risk of isolation and marginalization. The CRHESO project aims to analyze the factors influencing social functioning. The main hypothesis is that social functioning depends on various components, including neurocognitive, sociocognitive, and language abilities, along with their electrophysiological markers. CRHESO seeks to characterize neuropsychophysiological profiles (combining neuropsychological and electrophysiological data) to better understand social outcomes in individuals with schizophrenia and in healthy subjects.

The investigators will address the following objectives:

* Primary Objective: Primary Objective: To disentangle social functioning complexity in schizophrenia and healthy controls by characterizing neuropsychophysiological profiles linked to levels of social disruption
* Secondary Objective: To improve factors associated with social outcome and explore changes in neuropsychophysiological markers The investigators will enroll 50 schizophrenic patients and 50 healthy controls.

Participants will undergo an initial visit with a specialist psychiatrist who will verify that their conditions meet the criteria required by the study. Then, subjects will be tested for metaphor comprehension, as well as for the other variables included in the study, and the electrical brain activity will be registered through a 128 channel EEG.

To test if the factors associated with social dysfunction in schizophrenia can be restored, we will propose to subjects with schizophrenia to participate in a rehabilitative training. Those who choose not to undergo the training will only participate in the cross-sectional study, while 10 patients who decide to participate in the training will undergo cognitive remediation training (Cognitive Remediation), already published and demonstrated to be feasible for patients with schizophrenia.

In the check-up visits (i.e., after the training), the patients enrolled in the treatment group, will be tested for metaphor comprehension, as well as for the other variables included in the study, and the electrical brain activity will be registered through a 128 channel EEG.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Diagnosis of Schizophrenia according to DSM V criteria
* Ability to provide informed consent

Exclusion Criteria:

* Intellectual disability
* Neurological disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 subjects with schizopnrenia from San Raffaele Hospital (Milan) and 50 healthy controls living in Milan
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of the difference in neurocognitive data between patients and controls | through study completion, an average of 2.5 years
  Tracking down the alteration in neurocognitive abilities, evaluated with the Brief Assessment of Cognition in Schizophrenia (BACS) (standardized score 0-4)
Analysis of the difference in sociocognitive data between patients and controls | through study completion, an average of 2.5 years
  Tracking down the alteration in sociocognitive abilities, evaluated with the Picture sequencing task (PST) (score 0-56)
Analysis of the difference in pragmatic data between patients and controls | through study completion, an average of 2.5 years
  Tracking down the alteration in pragmatic abilities, evaluated with Assessment of Pragmatic Abilities and Cognitive Substrates (APACS brief) (score 0-1)
Analysis of the difference in language data between patients and controls | through study completion, an average of 2.5 years
  Tracking down the alteration in language abilities, evaluated with AWechsler Vocabulary task (score 0-66)
Tracking down the difficulties in metaphor comprehension via task during electrophysiological recording | through study completion, an average of 2.5 years
  Exploring the difference in the neurological correlates (via electrophysiological recording technique) between patients and controls. We will measure event-related potential (ERP) after the stimulus presentation
Analysis of the impact of neuropsychological and electrophysiological measures on quality of life | through study completion, an average of 2.5 years
  Evaluate the impact of neuropsychological and electrophysiological measures on quality of life, measured with the Quality of life scale (QLS) (score 0-126)
Analysis of the impact of neuropsychological and electrophysiological measures on community Integration | through study completion, an average of 2.5 years
  Evaluate the impact of neuropsychological and electrophysiological measures on community Integration, measured with the Community Integration measure (CIM) (score 10-50)
Analysis of the impact of neuropsychological and electrophysiological measures on social connectedness | through study completion, an average of 2.5 years
  Evaluate the impact of neuropsychological and electrophysiological measures on social connectedness, measured with the Social Connectedness scale (SCS-R) (score 20-120)

SECONDARY OUTCOMES:
Evaluation of psychopathology | through study completion, an average of 2.5 years
  Evaluate psychopathology with the Positive and Negative Syndrome scale (PANSS) (score 30-210)
Evaluate the efficacy of a rehabilitative training in restoring neurocognitive abilities | through study completion, an average of 2.5 years
  Test the improvement in neurocognitive abilities, evaluated with the Brief Assessment of Cognition in Schizophrenia (BACS) (standardized score 0-4)
Evaluate the efficacy of a rehabilitative training in restoring sociocognitive abilities | through study completion, an average of 2.5 years
  Test the improvement in sociocognitive abilities, evaluated with the Picture sequencing task (PST) (score 0-56)
Evaluate the efficacy of a rehabilitative training in restoring pragmatic abilities | through study completion, an average of 2.5 years
  Test the improvement in pragmatic abilities, evaluated with the Assessment of Pragmatic Abilities and Cognitive Substrates (APACS) (score 0-1)
Evaluate the efficacy of a rehabilitative training in restoring language abilities | through study completion, an average of 2.5 years
  Test the improvement in language abilities, evaluated with the Wechsler Vocabulary task (score 0-66)
Evaluate the efficacy of a rehabilitative training in restoring quality of life | through study completion, an average of 2.5 years
  Test the improvement of quality of life, measured with the Quality of life scale (QLS) (score 0-126)
Evaluate the efficacy of a rehabilitative training in restoring Community Integration | through study completion, an average of 2.5 years
  Test the improvement of Community Integration, measured with the Community Integration measure (CIM) (score 10-50)
Evaluate the efficacy of a rehabilitative training in restoring Social Connectedness | through study completion, an average of 2.5 years
  Test the improvement of Social Connectedness, measured with the Social Connectedness scale (SCS-R) (score 20-120)

IPD SHARING:
Plan to Share IPD: No